CLINICAL TRIAL: NCT07326514
Title: Electronic Real-Time Heart Team Decision-making vs. Usual Care in Patients With Triple-Vessel Coronary Artery Disease and Diabetes Mellitus
Acronym: EHEART-3VD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fuwai Yunnan Cardiovascular Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Central China Fuwai Hospital of Zhengzhou University (Other); Ruijin Hospital (Other); Nanjing First Hospital, Nanjing Medical University (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-2850
Record Dates: First submitted 2025-11-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Coronary Artery Disease
Keywords: coronary revascularization; heart team; implementation science
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time heart team group (Experimental): A online multidisciplinary heart team discussion and decision-making will be conducted during angiography
  Interventions: Other: Real-Time Heart Team Decision-making
- Usual care group (No Intervention): An usual care decision-making initiated by interventional cardiologists will be conducted

INTERVENTIONS:
Other: Real-Time Heart Team Decision-making — A online multidisciplinary heart team discussion and decision-making will be conducted during coronary angiography.
  Arms: Real-time heart team group

SUMMARY:
This is a multi-center randomized controlled trial involving patients with 3-vessel coronary artery disease and diabetes mellitus. Enrolled patients will be dividing into real-time heart team decision-making group (intervention group) and usual care group (control group). The intervention group will conduct a real-time online multidisciplinary heart team discussion and decision-making during coronary angiography. The control group will conduct an usual care decision-making.

ELIGIBILITY:
Inclusion Criteria (Fulfill 1,2,3 or 1,4):

1. Age ≥ 18 years;
2. Diabetes mellitus;
3. Three-vessel coronary artery disease (≥70% stenosis in the left anterior descending artery, circumflex artery, and right coronary artery system);
4. Patients who required heart team discussion judging by the interventional cardiologist.

Exclusion Criteria:

1. Prior PCI or CABG;
2. Acute myocardial infarction with ECG and biomarker tests indicating acute phase;
3. Concurrent severe valvular heart disease, large vessel disease, or giant ventricular aneurysm requiring surgical intervention;
4. Concurrent atrial fibrillation or severe arrhythmia;
5. Other emergency admissions where elective revascularization is contraindicated;
6. Refusal or rejection of a specific treatment options (PCI or CABG);
7. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
One-year composite of major adverse cardiac and cerebral events | 1 year
  One-year composite pf all-cause mortality, myocardial infarction, stroke, repeat revascularization, and rehospitalization for recurrent angina.

SECONDARY OUTCOMES:
Clinical adverse events | From randomization through 1-year follow-up (events recorded during index hospitalization and at follow-up visits up to 12 months).
  Incidence and time to first clinical event, including: all-cause mortality, cardiac mortality, non-fatal myocardial infarction, stroke, target-vessel or graft revascularization, repeat revascularization, unplanned revascularization, rehospitalization for recurrent angina, cardiac rehospitalization, and all-cause rehospitalization.
Guideline-concordant revascularization decision rate | During index hospitalization (typically within 30 days of admission)
  Proportion of coronary revascularization decisions that are concordant with the Guidelines class I or IIa recommendations.
Percutaneous coronary intervention (PCI) utilization rate | During index hospitalization (typically within 30 days of admission)
  Proportion of patients who undergo PCI as part of their coronary revascularization strategy.
Coronary artery bypass grafting (CABG) utilization rate | During index hospitalization (typically within 30 days of admission)
  Proportion of patients who undergo CABG as part of their coronary revascularization strategy.
Medical therapy rate | During index hospitalization (typically within 30 days of admission)
  Proportion of patients managed with medical therapy.
Waiting time from diagnostic angiography to treatment initiation | During index hospitalization (typically within 30 days of admission)
  Time from completion of diagnostic coronary angiography to initiation of the definitive treatment strategy (PCI, CABG, or medical therapy).
Medical costs | Index hospitalization until discharge (typically within 30 days of admission).
  Medical costs during the index hospitalization.
Hospital length of stay | From hospital admission to discharge for the index hospitalization (up to 30 days).
  Number of days from hospital admission to hospital discharge for the index hospitalization.
Prolonged PCI hospitalization | From index PCI procedure to discharge for the index hospitalization (up to 30 days).
  Proportion of patients with prolonged length of stay after PCI, defined according to the Centers for Medicare and Medicaid Services (CMS) criteria.
Time spent per heart team case | At the time of the heart team discussion during the index hospitalization (up to 30 days from admission).
  Duration of each heart team discussion.
Specialist satisfaction with discussion adequacy | Immediately after each heart team discussion during the index hospitalization (up to 30 days from admission).
  Satisfaction of participating specialists (interventional cardiologists and cardiac surgeons) with the adequacy of the discussion, assessed using a numeric rating scale (0-10, higher scores indicating greater satisfaction); reported as mean (±SD) score per group.
Seniority of participating specialist in heart team discussions | From index PCI procedure to discharge for the index hospitalization (up to 30 days)
  Proportion of specialists with different seniority, such as associated chief, chief etc..
Multidisciplinary synchronous shared decision-making | From index PCI procedure to discharge for the index hospitalization (up to 30 days)
  Proportion of cases in which interventional cardiology and cardiac surgery participate in a synchronous discussion with patient or relatives.
Patient satisfaction with the decision-making process | Within 24 hours before discharge from the index hospitalization (up to 30 days from admission).
  Patient-reported satisfaction with the coronary revascularization decision-making process, assessed using a structured questionnaire with a 5-point Likert scale.
Recatheterization rate | During index hospitalization (typically within 30 days of admission)
  Repeat invasive coronary angiography after the index procedure.
Specialist workload | During index hospitalization (typically within 30 days of admission)
  Workload of participating specialists based on NASA-TLX scale
Real-time consultation response rate | During index hospitalization (typically within 30 days of admission)
  A real-time response from cardiac surgeon during the coronary angiography.

IPD SHARING:
Plan to Share IPD: No